CLINICAL TRIAL: NCT04747093
Title: Induced-T Cell Like NK Cellular Immunotherapy for Refractory B Cell Malignancies
Brief Title: Induced-T Cell Like NK Cells for B Cell Malignancies
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Principal Investigator, Qifa Liu, Professor, Nanfang Hospital, Southern Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ITNK-2021
Record Dates: First submitted 2021-02-06; First posted 2021-02-10 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: B Cell Leukemia; B Cell Lymphoma; B-cell Acute Lymphoblastic Leukemia; B-cell Lymphoma Recurrent; B-cell Lymphoma Refractory
Keywords: ITNK Cells; CAR; B Cell Malignancy
MeSH Terms: conditions — Leukemia, B-Cell; Lymphoma, B-Cell; Burkitt Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ITNK group (Experimental)
  Interventions: Biological: CAR-ITNK cells

INTERVENTIONS:
Biological: CAR-ITNK cells — CAR-ITNK cells will be infused over 10-15 minutes on Day 0.

SUMMARY:
Relapsed and refractory B cell malignancies show unfavorable prognosis, especially for adult patients. Now, there is no standard management for these patients. Induced-T cell-like NK cells with chimeric antigen receptor (CAR-ITNK cells) is a promising treatment option for treating B cell derived malignancy. The purpose of this study is to evaluate the efficacy and safety of CAR-ITNK cells infusions in patients with relapsed and refractory B cell malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Patient with CD19 positive B-cell acute leukemia
* Eastern Cooperative Oncology Group (ECOG) performance status <2
* ALT/ AST <3 x normal
* Bilirubin < 2.0 mg/dl
* Creatinine < 2.5 mg/dl and less than 2.5x normal for age
* LVEF< 45%
* Accept white blood cell collection
* Provide informed consent

Exclusion Criteria:

* Previous treatment with investigational gene or cell therapy medicine products
* Active hepatitis B , hepatitis C or HIV infection
* Uncontrolled active infection
* Presence of grade 2-4 acute or extensive chronic GVHD
* Active CNS involvement: epilepsy, paresis, aphasia, stroke, severe head trauma,
* Dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, uncontrolled mental illness, etc.
* Any uncontrolled active medical disorder that would preclude participation as outlined.
* Received non-diagnostic purposes major surgery within the past 4 weeks
* Participated in any other clinical study within the past 4 weeks
* Used murine biological products (except blinatumomab), unless it is proved no anti-mouse antibodies exist.
* Pregnancy or breast-feeding women
* Use of prohibited drugs:
* Steroids: Therapeutic doses of steroids must be stopped > 72 hours prior to ITNK Cells infusion
* Allogeneic cellular therapy: Any donor lymphocyte infusions (DLI) must be completed > 4 weeks prior to ITNK Cells infusion
* GVHD therapies: Any drug used for GVHD must be stopped > 4 weeks prior to ITNK Cells infusion
* Any situation that may increase the risk of the test or interfere with the test results

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2021-01-29 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | 12 months

SECONDARY OUTCOMES:
ORR | 3 months
  Overall Response Rate includes Complete Remission (CR) and Complete Remission with Incomplete Blood Count Recovery (CRi), as determined by assessments of peripheral blood, bone marrow, CNS symptoms, physical exam (PE) and CSF. The primary endpoint will be based on the IRC assessment. The local investigator's assessed results will be used for sensitivity analysis.
ORR | 6 months
  Overall Response Rate includes Complete Remission (CR) and Complete Remission with Incomplete Blood Count Recovery (CRi), as determined by assessments of peripheral blood, bone marrow, CNS symptoms, physical exam (PE) and CSF. The primary endpoint will be based on the IRC assessment. The local investigator's assessed results will be used for sensitivity analysis.
ORR | 12 months
  Overall Response Rate includes Complete Remission (CR) and Complete Remission with Incomplete Blood Count Recovery (CRi), as determined by assessments of peripheral blood, bone marrow, CNS symptoms, physical exam (PE) and CSF. The primary endpoint will be based on the IRC assessment. The local investigator's assessed results will be used for sensitivity analysis.
OS | 1 year
  overall survival
DFS | 1 year
  disease-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Qi-fa Liu, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Department of Hematology,Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China